CLINICAL TRIAL: NCT01590160
Title: A Phase I/II Study of First Line Ganetespib With Platinum, in Patients With Malignant Pleural Mesothelioma
Brief Title: Ganetespib With Platinum, in Patients With Malignant Pleural Mesothelioma
Acronym: MESO-02
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0158; CMS # 1995 (Other Grant/Funding Number: Synta Pharmaceuticals); A15183 (Other Grant/Funding Number: Cancer Research UK Endorsement); 2012-001598-10 (EudraCT Number)
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer - Malignant Pleural Mesothelioma
MeSH Terms: interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin/Pemetrexed (Experimental): Cisplatin 75mg/m2, Day 1 every 21 days Pemetrexed 500mg/m2, Day 1 every 21 days
  Interventions: Drug: Ganetespib
- Carboplatin/Pemetrexed (Experimental): Carboplatin AUC5, Day 1 every 21 days Pemetrexed 500mg/m2, Day 1 every 21 days
  Interventions: Drug: Ganetespib

INTERVENTIONS:
Drug: Ganetespib — IV, Using dose from Phase I

SUMMARY:
Malignant pleural mesothelioma (MPM) is a rapidly lethal cancer arising from the parietal pleural mesothelium, and is associated with exposure to asbestos.

Once a rare disease, it is increasing in incidence in the UK and is presently more common than cervical cancer. MPM is characterized by local invasion of adjacent structures including the chest wall, mediastinum, diaphragm and pericardium resulting in progressive shortness of breath.

Median survival with best supportive care alone is approximately 6-9 months and most cases of mesothelioma present in the advanced setting. Therefore this trial will be looking at whether a new drug, Ganetespib has any improvement on survival for these types of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological confirmation of malignant pleural mesothelioma
2. Measurable disease using meso-modified RECIST criteria (CT scan must be within 28 days of registration/randomisation)
3. Performance status ECOG 0-1
4. Age at least 18 years
5. Adequate haematological status:

   * Haemoglobin 100g/L or greater
   * Neutrophil count ≥2.0 x 10^9/L
   * Platelets ≥100 x 10^9 /L
6. Adequate organ function:

   * Bilirubin ≤1.5x ULN, ALP ≤2.5x ULN, ALT or AST ≤1.5x ULN
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥ 60ml/min (C&G or EDTA)
7. Chemotherapy naïve
8. Negative serum pregnancy test for female patients of child bearing potential.
9. Male subjects and women of child bearing potential must agree to use an acceptable method of birth control for the duration of the trial and for 6 months after the last trial treatment cycle has finished.
10. Ability to understand and willing to sign the written informed consent to participate (including donation of diagnostic biopsy tissue for research)
11. Ability to comply with the requirements of the protocol

Exclusion Criteria:

1. Prior exposure to other investigational or commercial agents or therapies administered with the intent of treating the patient's malignancy. This includes crizotinib, other ALK-targeted agents, and any Hsp90 inhibitor (e.g. ganetespib). Prior valproic acid is acceptable but only if there has been at least 30 days wash-out period
2. Evidence of CNS metastases that in the opinion of the investigator should receive local treatment prior to systemic cytotoxic chemotherapy
3. Uncontrolled intercurrent illness including but not limited to:

   * Symptomatic neurological illness
   * Active uncontrolled systemic infection considered opportunistic, life threatening or clinically significant at the time of treatment
   * Significant pulmonary disease or hypoxia
   * Psychiatric illness/social situations that would limit compliance with trial requirements
   * Human immunodeficiency virus (HIV)-positive patients
   * Known hepatitis B or C infection
   * Uncontrolled diabetes mellitus
4. Serum potassium, magnesium, and calcium levels no more than 10% outside the Sites normal reference ranges
5. Known serious cardiac illness including but not confined to:

   * Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker
   * Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a Class Ia anti-arrhythmic drug (e.g., quinidine, procainamide, disopyramide) or Class III anti-arrhythmic drug (e.g., sotalol, amiodarone, dofetilide). Use of other anti-arrhythmic drugs is permitted.
   * Use of medications that have been linked to the occurrence of torsades de pointes
   * Second- or third-degree atrioventricular (AV) block unless treated with a permanent pacemaker
   * Complete left bundle branch block (LBBB)
   * History of long QT Syndrome or a family member with this condition
   * QTc >470ms (average of triplicate ECG recordings); a consistent method of QTc calculation must be used for each patient's QTc measurements. QTcF (Fridericia's formula) is preferred
6. The patient has a history of prior malignant tumour, unless the patient has been without evidence of disease for at least three years, or the tumour was a non-melanoma skin tumour or in situ cervix carcinoma
7. Pregnant women or those who are lactating
8. Pre-planned surgery or procedures that would interfere with the conduct of the trial
9. Patients who have had surgery (does not include pleurodesis or pleurectomy) within 28 days of randomisation should not be included
10. Previous treatment of mesothelioma with systemic chemotherapy
11. Receipt of extensive radiation therapy, systemic chemotherapy, or other anti-neoplastic therapy within 4 weeks before enrolment is not allowed. However, drain site radiotherapy is allowed
12. Significant weight loss (≥10% body weight) within the 4 weeks prior to Cycle 1 Day 1.
13. Patients who have had a yellow fever vaccination in the previous 30 days.
14. Other medications, severe acute/chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of Ganetespib | 6 Months
  Primary endpoint (phase I): Dose-limiting toxicities during Cycles 1 & 2; and number of cycles of pemetrexed-cisplatin given.
  The Phase I trial will consist of three ganetespib dose cohorts, each with 3 or 6 patients:
  * Cohort 1: 100mg/m2 IV on day 1 and day 15 of each cycle
  * Cohort 2: 150mg/m2 IV on day 1 and day 15 of each cycle
  * Cohort 3: 200mg/m2 IV on day 1 and day 15 of each cycle
  There will be additional patients to be treated with carboplatin (AUC5) instead of cisplatin. If treatment with carboplatin is confirmed to be safe and tolerable, the option of treating patients with either cisplatin or carboplatin during phase II will be taken. The evaluation will be done using an accelerated titrated phase I design.
  Primary endpoint (phase II): Progression free survival

SECONDARY OUTCOMES:
Progression Free Survival | 24 Months
  Secondary endpoints (phase I):
  * To examine the number of cycles of pemetrexed/platinum chemotherapy administered.
  * To examine the objective tumour response according to meso-modified RECIST, and the overall response rate.
  Secondary endpoints (phase II):
  * To examine the frequency of all Adverse Events graded by NCI-CTCAE version 4, in particular those with grade 3 or 4 events.
  * To examine the objective tumour response according to meso-modified RECIST, and the overall response rate.
  * To examine overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Professor D Fennell, MBBS, Study Chair — University of Leicester & Leicester University Hospitals
Locations (1):
- UCL Cancer Trials Centre, London, United Kingdom

REFERENCES:
- [Derived] Fennell DA, Danson S, Woll PJ, Forster M, Talbot D, Child J, Farrelly L, Sharkey A, Busacca S, Ngai Y, Hackshaw A, Wheeler GM. Ganetespib in Combination with Pemetrexed-Platinum Chemotherapy in Patients with Pleural Mesothelioma (MESO-02): A Phase Ib Trial. Clin Cancer Res. 2020 Sep 15;26(18):4748-4755. doi: 10.1158/1078-0432.CCR-20-1306. Epub 2020 Jul 15. PMID 32669375